CLINICAL TRIAL: NCT00643773
Title: The Influence of Leucine Supplementation on Body Composition and Muscle Characteristics in Elderly, Type 2 Diabetes Patients.
Brief Title: The Effect of Leucine on Body Composition and Muscle Characteristics in Elderly, Type 2 Diabetes Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Top Institute Food and Nutrition (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double
Other Study IDs: MEC-07-1111
Record Dates: First submitted 2008-03-20; First posted 2008-03-26 (Estimated); Last update posted 2011-08-26 (Estimated); Status verified 2011-08

CONDITIONS: Type 2 Diabetes
Keywords: Elderly
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Leucine; Flour

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Leucine supplement
  Interventions: Dietary Supplement: Leucine
- B (Placebo Comparator): Wheat flour
  Interventions: Dietary Supplement: Wheat flour

INTERVENTIONS:
Dietary Supplement: Leucine — capsules are 0.5g, subjects take 5 capsules with every main meal for 6 months In total this is 15 capsules per day
  Arms: A
Dietary Supplement: Wheat flour — Wheat flour
  Arms: B

SUMMARY:
The purpose of this study is to determine whether long term leucine supplementation has a positive effect on body composition and muscle characteristics in elderly, type 2 diabetes patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 2 diabetes

Exclusion Criteria:

* Impaired renal or liver function
* Cardiac disease
* Subjects with metal implants
* Hypertension
* Diabetes complications
* Exogenous insulin therapy

Min Age: 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-12 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Body Composition | 1, 3, and 6 months

SECONDARY OUTCOMES:
Muscle characteristics | 1, 3, and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Marika Leenders, MSc, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Netherlands

REFERENCES:
- [Derived] Leenders M, Verdijk LB, van der Hoeven L, van Kranenburg J, Hartgens F, Wodzig WK, Saris WH, van Loon LJ. Prolonged leucine supplementation does not augment muscle mass or affect glycemic control in elderly type 2 diabetic men. J Nutr. 2011 Jun;141(6):1070-6. doi: 10.3945/jn.111.138495. Epub 2011 Apr 27. PMID 21525248